CLINICAL TRIAL: NCT05289492
Title: Study of EOS884448 Alone, and in Combination with Iberdomide with or Without Dexamethasone, in Participants with Relapsed or Refractory Multiple Myeloma
Brief Title: Study of Novel Regimens in Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company operational decision. Decision to stop study is not due to safety or efficacy concerns
Sponsor: iTeos Therapeutics (Industry)
Collaborators: Bristol-Myers Squibb (Industry); GlaxoSmithKline (Industry); iTeos Belgium SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TIG-007
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; EOS884448; GSK4428859A; TIGIT; Anti-TIGIT; iberdomide; CELMoD; CC-220; EOS-448; Belrestotug
MeSH Terms: conditions — Multiple Myeloma | interventions — iberdomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- A: Participants will receive EOS884448 (Experimental): EOS884448 will be administered
  Interventions: Drug: EOS884448
- B: Participants will receive EOS884448 and iberdomide (Experimental): EOS884448 and iberdomide will be administered
  Interventions: Drug: EOS884448; Drug: Iberdomide
- C: Participants will receive EOS884448, iberdomide and dexamethasone (Experimental): EOS884448, iberdomide and dexamethasone will be administered
  Interventions: Drug: EOS884448; Drug: Iberdomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: EOS884448 — EOS884448 will be administered in arm A,B and C
  Other Names: EOS-448, GSK4428859A, Belrestotug
Drug: Iberdomide — Iberdomide will be administered in arm B and C
  Other Names: CC-220
  Arms: B: Participants will receive EOS884448 and iberdomide; C: Participants will receive EOS884448, iberdomide and dexamethasone
Drug: Dexamethasone — Dexamethasone will be administered in arm C
  Arms: C: Participants will receive EOS884448, iberdomide and dexamethasone

SUMMARY:
This is a multicenter, open-label, phase I/II clinical study, to assess the safety, tolerability, antitumor activity, pharmacokinetics and pharmacodynamics of EOS884448 (also known as EOS-448 or GSK4428859A), alone or in combination with iberdomide with and without dexamethasone in participants with relapsed/refractory multiple myeloma (RRMM).

ELIGIBILITY:
Inclusion Criteria:

* All participants must have a documented diagnosis of relapse/refractory Multiple Myeloma and have measurable disease as defined per IMWG criteria.
* All participants must have received at least 3 prior lines of MM therapy with IMiD, PI and Anti-CD-38, and progressed on their last therapy (prior BCMA targeted therapy allowed).
* All participants must have Eastern Cooperative Oncology Group (ECOG) Performance Status of 0,1or 2.
* All participants must have adequate organ function.
* Females of childbearing potential (FCBP) or male participant must agree to follow contraception requirements.

Exclusion Criteria:

* All participants with non-secretory MM
* All participants with known auto-immune disease
* All participants with history of life-threatening toxicity related to prior immune therapy.
* All participants with active graft versus host disease after allogeneic stem cell transplantation.
* All participants with active, unstable cardiovascular function.
* All participants with active infection requiring systemic therapy.
* All participants with hypersensitivity to any of the treatments.
* All participants with any active gastrointestinal dysfunction that prevents the patient from swallowing tablets or interferes with absorption of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Number of participants with any adverse events (AEs) and serious adverse events (SAEs) | From first study treatment administration up to 120 days after the last dose
Number of participants with dose limiting toxicity (DLT) | From first study treatment administration up to 120 days after the last dose
Recommended Phase 2 dose (RP2D) of EOS884448 alone or in combinations with iberdomide with or without dexamethasone in participants with relapse/refractory multiple myeloma | up to 2 years
Number of participants with overall response (partial or better) as determined by IMWG criteria | up to 2 years

SECONDARY OUTCOMES:
Progression-free-survival (PFS) | Until disease progression or death - Approximately 24 months
Duration of Response (DOR) | Until disease progression or death - Approximately 24 months
Time to Response (TTR) | Approximately 48 weeks
Maximum concentration (Cmax) of EOS884448 at each dose level | Approximately 48 weeks
Percentage of participants with anti-drug antibodies to EOS884448 | Approximately 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Iteos Clinical Trials, Study Director — iTeos Belgium SA
Locations (13):
- United States (4):
  - Banner MD Anderson, Gilbert, Arizona
  - Eastern Connecticut Hematology & Oncology, Norwich, Connecticut
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Belgium (3):
  - ZNA Cadix, Antwerp
  - Institut Jules Bordet, Brussels
  - Universitaire Ziekenhuizen KU Leuven, Leuven
- France (5):
  - CHU Amiens, Amiens
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - APHP Hôpital Saint-Antoine, Paris
  - CHU de Poitiers, Poitiers
  - CHU Toulouse, Toulouse
- Hospital Fundacion Jimenez Diaz, Madrid, Spain